CLINICAL TRIAL: NCT04449445
Title: Perioperative Nutritional Optimization in Head and Neck Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Barry Lloyd Wenig, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-1147
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard enteral tube feeds (Other): Patients will be instructed to continue a normal diet before surgery. Post-operatively, patients will receive standard of care isocaloric and iso-nitrogenous standard enteral tube feeds
  Interventions: Dietary Supplement: Isocaloric and iso-nitrogenous standard enteral tube feeds
- Nestle IMPACT AR (Experimental): Patients will be encouraged to continue their regular diet until their surgery day. In addition, beginning 5 days before surgery, subjects will be instructed to drink three, 6 ounce cartons of Nestle IMPACT AR each day until their surgery. Post operatively patients who are able to eat orally, will be given three, 6 ounce cartons of Nestle IMPACT AR to drink each day for 5 days. Patients who are not able to tolerate an oral diet will be given Nestle IMPACT via a continuous tube feeding for 5 days through a temporary nasogastric feeding tube placed per standard post-operative care. Dosing of the tube feeding will be based on weight at a rate of approximately 70-75 cc/hour.
  Interventions: Dietary Supplement: Nestle IMPACT AR

INTERVENTIONS:
Dietary Supplement: Isocaloric and iso-nitrogenous standard enteral tube feeds — Dietary supplement
  Arms: Standard enteral tube feeds
Dietary Supplement: Nestle IMPACT AR — Dietary supplement
  Arms: Nestle IMPACT AR

SUMMARY:
To determine whether nutritional optimization in head and neck cancer patients undergoing major surgery will decrease post-operative wound complications. The Investigators hypothesize that nutritional supplementation with Nestle Impact Advanced Recovery (AR) will decrease the rate of wound complications after surgery

DETAILED DESCRIPTION:
The purpose of this study is to determine whether nutritional optimization in head and neck cancer patients undergoing major surgery will decrease post-operative wound complications. It is likely that many head and neck cancer patients suffer from sarcopenia, and this contributes to many wound complications, including wound infection, dehiscence, fistula formation, and free flap tissue loss. The Investigators hypothesize that nutritional supplementation with Nestle Impact Advanced Recovery (AR) will decrease the rate of wound complications after surgery

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years. Both men and women and members of all races and ethnic groups will be included.
* Patients must be diagnosed with cancer of the head and neck and must be surgical candidates.
* Patients must be indicated for major head and neck surgery, defined as surgeries with an anticipated post-surgical hospital stay of 4 or more days. Examples of major surgeries include, but are not limited to, total laryngectomy, large oral cavity, oropharyngeal, salivary gland, or soft tissue resections requiring free flap or major regional flap (e.g. pectoralis major flap), and large skull base procedures requiring extensive skull base reconstruction.
* Patients must have cross-sectional body imaging (PET-CT or equivalent) performed within 4 weeks of study enrollment and available for review.
* Patient must be willing to receive Nestle IMPACT Advance Recovery for five days prior to planned surgery as well as for 5 days after surgery.
* Ability to understand and the willingness to sign a written informed consent document.
* All adult men and women with cancer of the head and neck undergoing surgery by the study PI's at UI Health will be considered for participation in this study without regard to race, gender or socioeconomic status.

Exclusion Criteria:

* Patients with known distant metastases or other malignancies.
* Patients unable to tolerate oral intake by mouth or per enteral feeding tube.
* Patients with galactosemia.
* Patients who have received any investigational medication within 6 weeks of enrollment, or who are scheduled to receive an investigational drug during the course of the study.
* Patients currently taking IMPACT or other immuno-nutrition products (arginine-containing supplements) will be excluded. Other forms of nutritional supplementation, such as caloric supplementation, tube feeding, or other dietary supplements are allowed on study.
* Patients currently taking anabolic steroids will be excluded. Patients taking corticosteroids are allowed on study.
* Psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of perioperative use of Nestle Impact AR | 30 days post-op
  Assess the rate of post-operative wound infection
Assess the effect of perioperative use of Nestle Impact AR | 30 days
  Assess the rate of post-operative seroma
Assess the effect of perioperative use of Nestle Impact AR | 30 days post-op
  Assess the rate of post-operative wound dehiscence
Assess the effect of perioperative use of Nestle Impact AR | 30 days post-op
  Assess the rate of post-operative fistula formation
Assess the effect of perioperative use of Nestle Impact AR | 30 days post-op
  Assess the rate of post-operative free tissue flap loss

SECONDARY OUTCOMES:
Assess whether sarcopenia is an independent risk factor for the development of post-operative wound complications | 30 days post-op
  A small biopsy of the sternocleidomastoid muscle will be taken to evaluate the presence of the key regulatory factors associated with sarcopenia
Assess whether sarcopenia is an independent risk factor for the development of post-operative wound complications | 30 days post-op
  Exome sequencing will be performed to assess expression of sarcopenia-related genes in peripheral blood
Assess whether sarcopenia is an independent risk factor for the development of post-operative wound complications | 30 days post-op
  Measurement of mean muscle mass at L3 on cross-sectional body imaging

CONTACTS AND LOCATIONS:
Overall Officials: Barry Wenig, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No